CLINICAL TRIAL: NCT05012644
Title: REAL-WORLD TUMOR RESPONSE OF PALBOCICLIB IN COMBINATION WITH AN AROMATASE INHIBITOR AS FIRST-LINE THERAPY IN PRE/PERIMENOPAUSAL WOMEN WITH METASTATIC BREAST CANCER
Brief Title: Comparative Real World Tumor Response in Pre-menopausal Metastatic Breast Cancer Patients Treated With Palbociclib + Aromatase Inhibitor or Aromatase Inhibitor Alone
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481159
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer
Keywords: pre-menopausal; palbociclib; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Palbociclib + aromatase inhibitor: Palbociclib + aromatase inhibitor
  Interventions: Drug: Palbociclib + aromatase inhibitor
- Aromatase inhibitor alone: Aromatase inhibitor alone
  Interventions: Drug: Aromatase inhibitor

INTERVENTIONS:
Drug: Palbociclib + aromatase inhibitor — Palbociclib + aromatase inhibitor
  Groups: Palbociclib + aromatase inhibitor
Drug: Aromatase inhibitor — Aromatase inhibitor
  Groups: Aromatase inhibitor alone

SUMMARY:
This study aims to assess real-world tumor response in pre/perimenopausal HR+/HER2- metastatic breast cancer (MBC) patients initiating palbociclib + aromatase inhibitor (AI) or AI alone as first-line therapy during the period on or after 01 January 2010 to on or before 30 June 2020. Data will be obtained from structured data fields within an electronic health record (EHR) database and will be supplemented by additional unstructured data collected through a targeted chart review.

ELIGIBILITY:
Inclusion Criteria:

1. Pre or perimenopausal at MBC diagnosis
2. Diagnosis of MBC in patient history
3. Confirmed HR+/HER2- status as defined as: a. HR+: ER+ or PR+ test; b. HER2-: any HER2 negative test and the absence of a positive test (IHC positive 3+, fluorescence in situ hybridization [FISH] positive/amplified, positive not otherwise specified [NOS]).
4. Received one of the following regimens as first-line treatment for MBC during the period from 01 January 2010 through index period 30 June 2020 until the data cutoff date of 31 December 2020.

   1. Palbociclib + AI as first-line treatment for MBC or
   2. Monotherapy AI as first-line treatment for MBC
5. Received care at a US Oncology Network (USON) site(s) utilizing the full EHR capacities of iKnowMed (iKM) at the time of treatment.
6. EHR data available from the USON site(s) where the patient received treatment are accessible for research purposes.

Exclusion Criteria:

1. Evidence of prior treatment with cyclin-dependent kinase (CDK) 4/6 inhibitors (palbociclib, ribociclib or abemaciclib) in the early breast cancer (BC) or MBC setting.
2. First structured activity (clinical visit) greater than 120 days after MBC diagnostic date with chart review to confirm no initial MBC treatment outside USON.
3. Receipt of treatment indicated for another primary cancer during the study observation period (after initiation of Palbociclib + AI or AI monotherapy and before 31 December 2020) or history of another primary cancer within USON.
4. Enrolled in any interventional clinical trial after initiation of Palbociclib + AI or AI monotherapy AND before 31 December 2020.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pre-menopausal metastatic breast cancer patients
Study Population: pre-menopausal metastatic breast cancer patients
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] DeMichele A, Robert N, Chen C, Kim S, Zhang Z, Lu DR, Aguilar KM, Wang Y, Li B, Schneeweiss S, Rassen JA, Gaffney M, McRoy L. Real-World Tumor Response of Palbociclib in Combination With an Aromatase Inhibitor as First-Line Therapy in Pre/Perimenopausal Women With Metastatic Breast Cancer. Target Oncol. 2023 Jul;18(4):543-558. doi: 10.1007/s11523-023-00979-1. Epub 2023 Jul 10. PMID 37428347
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from United States Oncology Network's (USON) iKnowMed (iKM) electronic health record (EHR) database combined with chart review in pre/perimenopausal patients with hormone receptor (HR) positive, human epidermal growth factor receptor (HER2) negative metastatic breast cancer (MBC) who initiated palbociclib plus aromatase inhibitor (AI) or AI alone as first-line therapy during the period of from 01 January 2010 to 30 June 2020 were assessed. The study data cutoff date was on 31 December 2020.
Pre-assignment Details: A total of 196 patients were included in the study, with 116 patients in the palbociclib plus AI cohort and 80 patients in the AI monotherapy cohort, after applying inclusion and exclusion criteria, using EHR structured data and chart review to confirm eligibility.
Groups:
- Palbociclib + AI: Pre/perimenopausal patients, diagnosed with HR positive (+), HER2 negative (-) MBC who initiated palbociclib along with AI as first-line therapy on or after 01 January 2010 up to and including 30 June 2020
- AI Monotherapy: Pre/perimenopausal patients, diagnosed with HR+, HER2- MBC who initiated AI alone as first-line therapy on or after 01 January 2010 up to and including 30 June 2020
Period: Overall Study
Arm/Group | Palbociclib + AI | AI Monotherapy
Started | 116 | 80
Discontinued (Included first line metastatic treatment only) | 64 | 67
Ongoing (Included first line metastatic treatment only) | 51 | 13
Completed (Included first line metastatic treatment only) | 1 | 0
Not Completed | 115 | 80

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Groups:
- Palbociclib + AI (All Patients): Patients who received palbociclib along with AI on or after 01 January 2010 up to and including 30 June 2020 for the treatment of MBC as part of their routine treatment were observed retrospectively.
- AI Monotherapy (All Patients): Patients who received AI alone on or after 01 January 2010 up to and including 30 June 2020 for the treatment of MBC as part of their routine treatment were observed retrospectively.
- Total: Total of all reporting groups
Arm/Group | Palbociclib + AI (All Patients) | AI Monotherapy (All Patients) | Total
Number analyzed (Participants) | 116 | 80 | 196
Age, Customized [Count of Participants; unit: Participants]
  <30 Years | 2 | 0 | 2
  30-44 Years | 45 | 29 | 74
  >=45 Years | 69 | 51 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 80 | 196
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 14 | 9 | 23
  White | 76 | 55 | 131
  Not Reported | 19 | 12 | 31
  Unknown | 7 | 4 | 11
Body Mass Index (BMI) (>= 25) [Count of Participants; unit: Participants]
  Yes | 75 | 41 | 116
  No | 33 | 26 | 59
  Unknown | 8 | 13 | 21
Disease Site (s) [Count of Participants; unit: Participants]
  Visceral | 43 | 29 | 72
  Non-visceral | 42 | 17 | 59
  Bone Only | 31 | 34 | 65
Number of Metastatic Site(s) [Count of Participants; unit: Participants]
  1 | 31 | 30 | 61
  2 | 42 | 20 | 62
  3+ | 43 | 30 | 73
Stage at Diagnosis [Count of Participants; unit: Participants] — Stage refers to the extent of your cancer, such as how large the tumor is and if it has spread. Stage is determined by X-rays, lab tests and other tests or procedures. Tumor, Node, Metastasis (TNM) combinations were used. TNM combinations were grouped into 5 stages: Stage 0 = abnormal cells were present but had not spread to nearby tissue; Stage I, Stage II and Stage III = Cancer was present. The higher the number, the larger the cancer tumor and the more it had spread into nearby tissues; Stage IV = The cancer has spread to distant parts of the body.
  Participants
    Stage 0 | 1 | 0 | 1
    Stage I | 21 | 9 | 30
    Stage II | 38 | 26 | 64
    Stage III | 21 | 21 | 42
    Stage IV | 30 | 20 | 50
    Unknown | 5 | 4 | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG performance status score is a rating of a patient's disease status, daily living activities and quality of life, with low scores indicating greater functioning than high scores: 0 = fully active; 1 = restricted in physically strenuous; 2 = ambulatory and capable of self-care but unable to work; 3 = capable of self-care but unable to work; 4 = completely disabled; 5 = dead. 2+ included those participants with ECOG performance status scores of 2-5.
  Participants
    0 | 34 | 27 | 61
    1 | 42 | 24 | 66
    2+ | 8 | 9 | 17
    Unknown | 32 | 20 | 52
Prior Neo/Adjuvant Chemotherapy [Count of Participants; unit: Participants]
  Yes | 50 | 36 | 86
  No | 66 | 44 | 110
Disease-free Interval [Count of Participants; unit: Participants]
  < 12 Months | 54 | 32 | 86
  >= 12 Months | 14 | 18 | 32
  De Novo Metastatic | 35 | 22 | 57
  Unknown | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Real World Tumor Response (rwTR) of All Participants (Adjusted by Normalized Inverse Probability of Treatment Weighting [nIPTW])
Description: rwTR of complete response (CR) or partial response (PR) based on response assessments captured with chart review during first line therapy. Real-world response rate (rwRR) was estimated using nIPTW method to adjust for the potential imbalance between the 2 treatment cohorts. CR was documented as 'a complete response' to therapy, indication patient is in 'remission', 'all lesions' have disappeared, or 'no evidence of disease'. PR was documented as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease (decrease in disease volume even though disease is still present). nIPTW method was employed to reduce confounding due to potential selection biases.
Time Frame: 11 Years. From 01 January 2010 to 30 June 2020 were assessed. The study data cutoff date was on 31 December 2020.
Population: Pre/perimenopausal patients who were treated with palbociclib plus AI or AI monotherapy as first-line treatment for HR positive, HER2 negative MBC in the US clinical practice setting from the USON database who met the inclusion/exclusion criteria of the study protocol. The study period began at patients' starting date of the first-line MBC treatment during the period of 01 January 2010 through 30 June 2020 to study end (data cutoff 31 December 2020).
Measure: Number; unit: Percentage of Participants
Groups:
- Palbociclib + AI: Patients who received palbociclib along with AI on or after 01 January 2010 up to and including 30 June 2020 for the treatment of MBC as part of their routine treatment were observed retrospectively. Normalized inverse probability of treatment weighting (nIPTW) adjustment was applied.
- AI Monotherapy: Patients who received AI alone on or after 01 January 2010 up to and including 30 June 2020 for the treatment of MBC as part of their routine treatment were observed retrospectively. Normalized inverse probability of treatment weighting (nIPTW) adjustment was applied.
Arm/Group | Palbociclib + AI | AI Monotherapy
Number analyzed (Participants) | 116 | 80
Percentage of Participants | 52.1 | 46.2
Statistical Analysis 1: Comparison: Palbociclib + AI vs AI Monotherapy; Test type: Other; Odds Ratio (OR) = 1.266, 95% CI 2-sided [0.715 to 2.241]

2. Primary Outcome: Real World Tumor Response in Patients With Tumor Assessment (Adjusted by nIPTW)
Description: rwTR of complete CR or PR based on response assessments captured with chart review during first line therapy. rwRR was estimated using nIPTW method to adjust for the potential imbalance between the 2 treatment cohorts. CR was documented as 'a complete response' to therapy, indication patient is in 'remission', 'all lesions' have disappeared, or 'no evidence of disease'. PR was documented as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease (decrease in disease volume even though disease is still present). nIPTW method was employed to reduce confounding due to potential selection biases.
Time Frame: 11 Years. From 01 January 2010 to 30 June 2020 were assessed. The study data cutoff date was on 31 December 2020.
Population: A subgroup of patients with at least 1 tumor assessment on treatment, from pre/perimenopausal patients treated with palbociclib plus AI or AI monotherapy as first-line treatment for HR positive, HER2 negative MBC in the US clinical practice setting from the USON database who met the eligibility of the study protocol. Began at patients' starting date of the first-line MBC treatment from 01 January 2010 to 30 June 2020 to study end (data cutoff 31 December 2020).
Measure: Number; unit: Percentage of Participants
Arm/Group | Palbociclib + AI | AI Monotherapy
Number analyzed (Participants) | 103 | 71
Percentage of Participants | 60.0 | 49.9
Statistical Analysis 1: Comparison: Palbociclib + AI vs AI Monotherapy; Test type: Other; Odds Ratio (OR) = 1.508, 95% CI 2-sided [0.819 to 2.774]

ADVERSE EVENTS:
Time Frame: 11 Years.
Description: Due to non-interventional nature of the study, safety data was collected as standard non-interventional study reporting only, with the exception of for ILD and pneumonitis.
Arm/Group | Palbociclib + AI | AI Monotherapy
All-Cause Mortality (participants affected / at risk) | 27/116 | 38/80
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/80
Other Adverse Events (participants affected / at risk) | 0/116 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05012644/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT05012644/SAP_001.pdf